CLINICAL TRIAL: NCT05376306
Title: Effects of Stress Management Interventions on STEM and Non-STEM Students
Brief Title: Stress Interventions in STEM and Non-STEM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Andrea M. Spaeth, PhD, Assistant Professor, Undergraduate Academic Director, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021001528
Record Dates: First submitted 2022-03-16; First posted 2022-05-17 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: MBSR-STEM; PMR-STEM; MBSR-NON-STEM; PMR -NON-STEM
Keywords: stress; sleep; STEM; non-STEM; students; stress interventions; PMR; MBSR
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MBSR - STEM (Experimental): STEM MAJOR in COLLEGE randomized to receive Mindfulness-based Stress Reduction intervention
  Interventions: Behavioral: Stress Reduction: MBSR
- MBSR - non-STEM (Experimental): Non-STEM MAJOR in COLLEGE randomized to receive Mindfulness-based Stress Reduction intervention
  Interventions: Behavioral: Stress Reduction: MBSR
- PMR - STEM (Experimental): STEM MAJOR in COLLEGE randomized to receive Progressive Muscle Relaxation intervention
  Interventions: Behavioral: Stress Reduction : PMR
- PMR - Non-STEM (Experimental): Non-STEM MAJOR in COLLEGE randomized to receive Progressive Muscle Relaxation intervention
  Interventions: Behavioral: Stress Reduction : PMR

INTERVENTIONS:
Behavioral: Stress Reduction: MBSR — Four activities, one each week - raising body awareness, sitting meditation, mindful yoga, expanding awareness meditation.
  Arms: MBSR - STEM; MBSR - non-STEM
Behavioral: Stress Reduction : PMR — Progressively tensing and releasing each muscle group from head to toe in a specific order.
  Arms: PMR - Non-STEM; PMR - STEM

SUMMARY:
The purpose of this study is to determine if (1) stress management intervention response depends on college major and (2) if there is a difference in effectiveness between Mindfulness Based Stress Reduction (MBSR) and Progressive Muscle Relaxation (PMR).

A. Objectives The goal of this study is to determine if STEM and non-STEM students respond differently to stress management interventions (SMIs) and to measure if MBSR and PMR are effective for reducing stress and improving sleep, mood, anxiety and depression symptoms.

B. Research Question(s) Aim #1: Determine if the type of SMI (PMR or MBSR) has different efficacies on STEM vs nonSTEM students for reducing stress and improving sleep, mood, anxiety and depression in university students.

Aim #2: Determine if administration of a SMI improves self-reported stress, sleep quality, mood, anxiety and depression in university students.

DETAILED DESCRIPTION:
Stress is a common response throughout all populations but has been associated with a 20% increase in the last thirty years. There are positive aspects to stress but high levels of consistent stress can be detrimental on the individual. In 2014, 77% of all Americans reported regularly experiencing physical symptoms of stress and 73% reported regularly experiencing the psychological effects caused by stress, with 33% feeling that they are dealing with extreme stress. When stress levels remain high for prolonged periods of time, individuals can experience the risk of development or worsening of sleep issues. There is abundant evidence that stress can cause changes in sleep time, fragmented sleep patterns, time taken to fall asleep, etc. Dysregulation of sleep is associated with worsening and development of mental health disorders like anxiety and depression. Stress can also adversely impact health due to its effect on suppressing the immune system and has a major impact on the severity of negative moods in individuals.

College students are a subset of the population that are vulnerable to experiencing extreme and prolonged stress, and in turn, poor sleep quality and depressive and anxiety symptoms. College students are a unique population as they are living in a critical period experiencing major environmental and psychological challenges and adaptations. Nearly 60% of all college students are reporting facing higher than average stress which is at an all-time high. College students already report poor sleep hygiene and quality which makes the impact of stress more profound on their health. Depressive symptoms across universities worldwide show that up to 50% of college students are facing depressive symptoms regularly. In a separate study, it was found that 3 out of 4 American college students in 2017 have experienced a sense of overwhelming anxiety. There is also a strong association with self-reported low sleep quality and experience of depression or depressive symptoms and anxiety symptoms, indicating the high levels of stress in college students are indirectly responsible for mental health concerns.

Stress in college students has become more prevalent in the past year due to the COVID-19 pandemic which resulted in many students living at home and having a virtual education. In 2020, individuals aged 18-23 (Gen Z adults) were reported as having the highest stress levels compared to other age groups. 87% of Gen Z adults in college reported that education and uncertainty about academics due to the COVID-19 pandemic were the reason for the higher stress levels. Gen Z adults were also most likely to report depressive symptoms with 34% saying that their mental health was worse than the prior year. In a separate study, sleep patterns in 86% of college students during the pandemic were shown to have been severely disrupted. Increased stress as a consequence of the pandemic has had direct effects on stress which has in turn deteriorated sleep quality and the mental health of college age kids.

Efforts to reduce stress in college age kids have been studied in the past. One such study looks at the efficacy of using a mindfulness meditation mobile app which was shown to reduce stress and improve sleep disturbances. Mindfulness, cognitive, and behavioral intervention programs have also been administered with evidence that they can be effective in stress reduction in college students. Prior studies have tested the effects of stress reduction interventions on a general college student population without taking into account differences within the types of stress that college students face. A major contributor to stress for college students is the major they choose- specifically whether the student chooses a STEM major or a non-STEM major. STEM majors consist of the most stressful fields of study according to Indiana University's National 2016 Study of Student Engagement. Self-reported scores of stress were the highest among STEM students and STEM students were also more likely to pull more all-nighters, have more homework, and less sleep compared to humanities majors. STEM majors also report studying and preparing the most number of hours compared to other majors.

STEM students also differ from non-STEM students with regards to engagement with their institution. Non-STEM college students displayed higher integrative and learning skills and scored higher on Higher Order Thinking surveys compared to STEM students. These differences in cognitive behaviors could result in stress interventions that require deeper reflection like Mental Imagery and Mindfulness Interventions to be more effective in non-STEM students than in STEM students. Understanding these differences in how STEM and non-STEM students respond to different stress interventions can allow students and universities to help alleviate the adverse effects of stress.

ELIGIBILITY:
Inclusion Criteria:

* They must be a current Rutgers University undergraduate student
* They are between the ages of 18 and 23
* They must have a declared major o They must be English speaking
* They must be able to comprehend all procedures and measures
* They are willing to complete all study procedures including the 6 week SMI

Exclusion Criteria:

* They currently have or have a history of sleep apnea
* They are a double major, with one major in STEM and the other in non-STEM

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Self Reported Stress | up to study completion, average of 1 month
  The Perceived Stress Questionnaire (PSQ) is used to determine a patient's subjective perceived stress.

SECONDARY OUTCOMES:
Anxiety Symptoms | Pre and post intervention (up to study completion, average of 1 month)
  The Beck Anxiety Inventory (BIA) is used to assess self-reported anxiety symptoms.
Depressive Symptoms | Pre and post intervention (up to study completion, average of 1 month)
  The Beck Depression Inventory (BDI) is designed to evaluate the severity of depression in normal and psychiatric populations.
Sleep quality | Pre and post intervention (up to study completion, average of 1 month)
  The Sleep Quality Scale (SQS) is used to measure sleep quality.
Sleep quality | Pre and post intervention (up to study completion, average of 1 month)
  The Pittsburgh Sleep Quality Index (PSQI) is used to measure sleep quality.
Mood | Pre and post intervention (up to study completion, average of 1 month)
  The Abbreviated Profile of Mood States is used to assess self-reported mood states.
Sleep Hygiene | Pre and post intervention (up to study completion, average of 1 month)
  The Sleep Hygiene Index (SHI) was used to measure self-reported sleep hygiene.

CONTACTS AND LOCATIONS:
Overall Officials: Pranav Reddy, Study Director — Rutgers University, Department of Kinesiology and Health -; Andrea Spaeth, PhD, Principal Investigator — Rutgers University, Department of Kinesiology and Health -
Locations (1):
- Rutgers Sleep Lab, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/23246209/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24965313/
- See also: Related Info — http://www.apa.org/news/press/releases/stress/2017/state-nation.pdf
- See also: Related Info — http://www.apa.org/news/press/releases/stress/2020/report-october
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5110386
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3586742
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/3204199/
- See also: Related Info — http://link.springer.com/article/10.1007/s12671-014-0356-5
- See also: Related Info — https://hqlo.biomedcentral.com/articles/10.1186/1477-7525-11-213#:~:text=The%20NRS%20has%20been%20shown%20to%20have%20adequate,scale%20ra%20nging%20from%200%20%28never%29%20to%204%20%28always%29
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6361309/
- See also: Related Info — https://eric.ed.gov/?id=EJ1191144
- See also: Related Info — http://www.semanticscholar.org/paper/Effectiveness-of-Progressive-Muscle-Relaxation-on-Gangadharan-Madani/ea750e4c6fbe58ce154eb68845d7d2c29e533426
- See also: Related Info — https://www.researchgate.net/publication/232536671_Preliminary_evidence_for_the_reliability_and_validity_of_an_abbreviated_Profile_of_Mood_States
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/15673628/
- See also: Related Info — https://www.semanticscholar.org/paper/Manual-for-the-Profile-of-Mood-States-Mcnair-Lorr/4d52b575f9055d62903bc0b829c1da475f5d571f
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2215737/
- See also: Related Info — https://scholarship.shu.edu/cgi/viewcontent.cgi?article=3687&context=dissertations
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9636945/
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2568977/
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC7473764/
- See also: Related Info — https://connect.springerpub.com/content/sgrrrpe/32/4/232
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/16911033/